CLINICAL TRIAL: NCT05964686
Title: The Efficacy of 2780 nm Er,Cr;YSGG and 940 nm Diode Laser in Root Canal Disinfection: A Randomized Clinical Trial
Brief Title: The Efficacy of Laser in Root Canal Disinfection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Zakaria Fahim, assistant lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID 041908
Record Dates: First submitted 2023-07-04; First posted 2023-07-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-07

CONDITIONS: Pulp and Periapical Tissue Disease; Pulp Necroses; Pulp; Granuloma
Keywords: LASER; Endodontics; canal disinfection
MeSH Terms: conditions — Dental Pulp Necrosis; Granuloma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional group A (Active Comparator)
  Interventions: Combination Product: Conventional group (NaOCl/EDTA)
- Dual laser group B (Experimental)
  Interventions: Combination Product: Dual laser group (Er,Cr:YSGG/Diode):
- Combined group C (Experimental)
  Interventions: Combination Product: Combined group (EDTA/Diode):

INTERVENTIONS:
Combination Product: Conventional group (NaOCl/EDTA) — conventional disinfection using 2.5% sodium hypochlorite and 17% EDTA
  Arms: Conventional group A
Combination Product: Dual laser group (Er,Cr:YSGG/Diode): — Er,Cr:YSGG intracanal laser irradiation to remove smear layer followed by diode laser for disinfection
  Arms: Dual laser group B
Combination Product: Combined group (EDTA/Diode): — 17% EDTA was used to remove smear layer followed by diode laser for disinfection
  Arms: Combined group C

SUMMARY:
The aim of this study is to assess in vivo the efficacy of Er,Cr:YSGG/diode laser and Diode/EDTA on bacterial count in root canal treatment in an evidence-based clinical trial. The null hypothesis being tested is that there is no difference in total bacterial count reduction between conventional irrigation and the two types of lasers used.

Thirty patients are equally divided into 3 separate groups :

* Group A (Conventional): 2.5% NaOCL and 17% EDTA.
* Group B(Dual): saline along with Er,Cr:YSGG laser and diode laser combination
* Group C(Combined): saline along with 17% EDTA and diode laser combination Microbiological analysis will be done for both aerobic and anaerobic bacteria using Colony forming units. All data will be collected, tabulated, summarized, and statistically analyzed.

DETAILED DESCRIPTION:
The use of lasers in disinfection of the root canal has been recently implemented. Lasers have bactericidal effect, and have deep penetration depth inside the root canal up to 1000 um. Thus, it can be used effectively for disinfection of the root canal system following biomechanical instrumentation reaching areas which were considered before non-reachable.

The aim of this study is to assess in vivo the efficacy of Er,Cr:YSGG/diode laser and Diode/EDTA on root canal treatment in an evidence-based clinical trial. The null hypothesis being tested is that there is no difference in total bacterial count reduction between conventional irrigation and the two types of lasers used.

Thirty patients are equally divided into 3 separate groups :

* Group A (Conventional): 2.5% NaOCL and 17% EDTA.
* Group B(Dual): saline along with Er,Cr:YSGG laser and diode laser combination
* Group C(Combined): saline along with 17% EDTA and diode laser combination After disinfection, local anesthetic and tooth isolation and access cavity preparation, the first microbial samples (S1) will be collected using 3 sterile paper points and immediately placed inside sterile tubes containing transport medium of thioglycolate, cleaning and shaping with final disinfection protocol will be performed according to the group in which the participant was allocated to. Followed by S2 sample. obturation using warm vertical compaction technique. Microbiological analysis will be done for both aerobic and anaerobic bacteria using Colony forming units. All data will be collected, tabulated, summarized, and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are medically free.

  * Patient's age between 18-35 years.
  * One single rooted maxillary anterior tooth with necrotic pulp and asymptomatic apical periodontitis requiring root canal treatment.
  * Patients complaining of no pain and without fistulous tract.
  * Periapical lesion with a periapical index score of 3 or 4 (Ørstavik, et al. (1986)108
  * Closed apex.
  * Acceptance to participate in the study.

Exclusion Criteria:

* Patients suffering from any systemic disease.
* Patients who had received antibiotics during the last month.
* Patients taking analgesics 12 hours before interventions.
* Patients with history of tobacco usage
* Teeth with vital pulp, calcified canals, and immature or incompletely formed apices.
* Teeth with previous endodontic treatment.
* Non restorable teeth where rubber dam could not be applied.
* Teeth with periodontal pocket more than 3 mm.
* Teeth with greater than grade 1 mobility.
* Teeth with swelling/sinus tract.
* Technical difficulties in the course of root canal treatment for example:

  * A tooth with curved roots

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Quantitative microbiological analysis | baseline (S1): sample will be obtained before canal disinfection. post operative (S2): sample will be obtained after canal disinfection in a single visit]
  aerobic bacterial count will be assessed using colony forming units (CFU) and will be expressed in (CFU/ml).
  anaerobic bacterial count will be assessed using colony forming units (CFU) and will be expressed in (CFU/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt